CLINICAL TRIAL: NCT03394677
Title: Phase 2 Study to Evaluate the Efficacy, Safety, and Tolerabililty of RVT-501 Topical Ointment in Pediatric Patients With Mild to Moderate Atopic Dermatitis
Brief Title: Study of RVT-501 Topical Ointment in Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dermavant Sciences GmbH (Industry)
Responsible Party: Sponsor
Organization: Dermavant Sciences, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-501-2004
Record Dates: First submitted 2017-12-21; First posted 2018-01-09 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — methyl 4-(((3-(6,7-dimethoxy-2-(methylamino)quinazolin-4-yl)phenyl)amino)carbonyl)benzoate; Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RVT-501 0.5% ointment (Experimental): Subjects will receive RVT-501 0.5% ointment twice daily (BID) for 4 weeks.
  Interventions: Drug: RVT-501 0.5% ointment
- RVT-501 vehicle ointment (Placebo Comparator): Subjects will receive RVT-501 vehicle ointment twice daily (BID) for 4 weeks.
  Interventions: Drug: Vehicle ointment

INTERVENTIONS:
Drug: RVT-501 0.5% ointment — Patients will receive RVT-501 0.5% ointment twice daily (BID) for 4 weeks.
  Arms: RVT-501 0.5% ointment
Drug: Vehicle ointment — Placebo comparator - ointment twice daily (BID) for 4 weeks.
  Arms: RVT-501 vehicle ointment

SUMMARY:
This is a multi-center, randomized, vehicle controlled, double-blind Phase 2 study in pediatric patients age 2-17 years old with mild to moderate atopic dermatitis.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, efficacy, and tolerability of a 0.5% BID concentration of RVT-501 in pediatric patients 2-17 years of age with mild to moderate atopic dermatitis. The pharmacokinetics of RVT-501 will also be evaluated in patients 2-11 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female pediatric patients ages 2-17 years of age with confirmed diagnosis of atopic dermatitis by Hanifin and Rajka criteria [Hanifin, 1980].
2. Patients with atopic dermatitis covering 5% to 40% of the body surface area (BSA) and with an Investigator Global Assessment (IGA) of 2 or 3 (mild or moderate atopic dermatitis) at Baseline. Scalp, palms, and soles should be excluded from the BSA calculation to determine eligibility at Baseline.

   Note: Patients with mild disease (IGA = 2) will be limited to approximately 25% of total enrollment.
3. Females of childbearing potential and male patients who are engaging in sexual activity that could lead to pregnancy must use the following adequate birth control methods while on study and for 2 weeks after stopping the study drug. Acceptable contraception methods are:

   * Male or male partner with vasectomy, OR
   * Male condom AND partner use of one of the contraceptive options below:
   * Spermicide;
   * Contraceptive subdermal implant that meets effectiveness criteria including a <1% rate of failure per year, as stated in the product label;
   * Intrauterine device or intrauterine system that meets effectiveness criteria including <1% rate of failure per year, as stated in the product label;
   * Oral contraceptive, either combined or progestogen alone;
   * Injectable progestogen;
   * Contraceptive vaginal ring;
   * Percutaneous contraceptive patches.

   These allowed methods of contraception are only effective when used consistently, correctly, and in accordance with the product label. The Investigator is responsible for ensuring that patients understand how to properly use these methods of contraception.

   Non-child-bearing potential is defined as pre-menarchal or pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy (removal of the ovaries) or hysterectomy, or hysteroscopic sterilization. Documented verbal history from the patient is acceptable.

   Patients who are abstinent are eligible, but they must agree to use of one of the birth control methods listed above if they start engaging in sexual activity that could lead to pregnancy during the study.

   Female subjects of childbearing potential must have a negative pregnancy test at Screening and Baseline (Day 0).
4. History of atopic dermatitis and stable disease for at least 1 month according to the patient/caregiver.
5. Patient, patient's parent(s), or legal representative must be capable of giving written informed consent or verbal assent, as applicable, which includes compliance with the requirements and restrictions listed in the consent/assent form; written informed consent must be obtained prior to any study related procedures.

Exclusion Criteria:

1. A positive Hepatitis B surface antigen (HBsAg) or positive Hepatitis C antibody result, or positive human immunodeficiency virus (HIV) antibody at Screening.
2. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 1.5x the upper limit of normal (ULN).
3. Screening total bilirubin > 1.5x ULN; total bilirubin > ULN and ≤ 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%.
4. Patients with a skin condition such as Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo, psoriasis, severe acne, connective tissue disorder, or Netherton's syndrome, or any other disease that could impact study evaluations.
5. Use of any prohibited medication.

   Prohibited concomitant medications, therapy, etc. during the defined period are as listed in the bullets below. If a patient requires any of these medications throughout the study period, he/she may be excluded from or discontinued from the study, at the discretion of the Investigator and medical monitor.

   - From 6 months prior to the first application of study drugs to the completion of the

   Follow-up visit or discontinuation:
   * Biological products that might have significantly affected the evaluation of atopic dermatitis condition (e.g., tumor necrosis factor [TNF] inhibitors, anti- immunoglobulin [Ig]E antibodies, anti-CD20 antibodies, anti-interleukin [IL]-4 receptor).
   * From 28 days prior to the first application of study drug until the completion of the Follow- up visit or discontinuation:
   * Corticosteroid preparations (oral, injection, and suppository preparations) and topical corticosteroids that were classified as super-high potency (clobetasol propionate). Eye drop and nasal preparations are allowed. Inhaled preparations are allowed if used for a stable condition and at a stable dose for > 28 days before Screening, and are continued at the same dose throughout the study.
   * Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, etc.);
   * Excessive sun exposure, tanning booth, other ultraviolet (UV) light source and phototherapy including psoralen and ultraviolet A (PUVA) therapy.
   * From 14 days prior to the first application of the study drug to the completion of the

   Follow-up visit or discontinuation:
   * Herbal medicines for atopic dermatitis (topical and oral preparations), unless specifically approved by the sponsor;
   * Eucrisa™ (crisaborole) and any other topical phosphodiesterase 4 (PDE4) inhibitor;
   * Tacrolimus and pimecrolimus cream and/or ointment;
   * Topical corticosteroids that were classified as low, medium, or high potency (fluocinonide, triamcinolone acetonide, desonide, hydrocortisone). Eye drops and nasal preparations are allowed.
   * From 7 days prior to the first application of the study drug to the completion of the

   Follow-up visit or discontinuation:
   * Oral or intravenous antibiotics, antifungal or antivirus medications
   * Antihistamines/anti-allergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine).

   NOTE: The following antihistamines are allowed:
   * Loratadine, fexofenadine hydrochloride, cetirizine hydrochloride
6. Pregnant or lactating females.
7. History of sensitivity to the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or medical monitor, contraindicates their participation.
8. The patient has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is longer).
9. Current or a history of cancer within 5 years.
10. Patients with active infection in atopic dermatitis areas requiring antibiotics, antifungals, or antiviral agents within 7 days of Baseline (Day 0).
11. Patients with pruritus due to conditions other than atopic dermatitis that, in the opinion of the Investigator, would either interfere with study evaluations or affect the safety of the patient.
12. Patients with advanced disease or recent abnormal laboratory test values that could affect the safety of the patient or the implementation of this study, as determined by medical records.
13. History of and/or concurrent condition of serious hypersensitivity (anaphylactic shock or anaphylactoid reaction) to PDE4 inhibitors.
14. Prior exposure to RVT-501.
15. Evidence of significant hepatic, renal, respiratory, endocrine, hematologic, neurologic, psychiatric, or cardiovascular system abnormalities or laboratory abnormalities that will affect the health of the patient or interfere with interpretation of the results.
16. The patient has excessive sun exposure, is planning a trip to a sunny climate that would involve excessive sun exposure, or used tanning booths within 28 days prior to Baseline (Day 0) or is not willing to minimize natural and artificial sunlight exposure during the study.

Other Eligibility Criteria Considerations:

To assess any potential impact on patient eligibility with regard to safety, the Investigator must refer to the following document for detailed information regarding warnings, precaustions, contraindications, adverse events, and other significant data pertaining to the investigational product being used in the study:

* The current version of the RVT-501 Investigator's Brochure.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Efficacy - Investigator Global Assessment (IGA) score | 28 days
  Efficacy will be assessed by determining the proportion of patients who achieve an Investigator Global Assessment (IGA) score of 0 or 1 and at least a 2-point improvement in IGA at Week 4. The IGA will be assessed at every study visit. The IGA is a 5-point morphological assessment of overall disease severity and will be determined according to the following categories: 0-clear; 1-almost clear; 2-mild disease; 3-moderate disease; 4-severe disease.
Efficacy - Eczema Area Severity Index (EASI) score | 28 days
  Efficacy will be assessed by determining the proportion of patients who achieve a 50% reduction in Eczema Area Severity Index score (EASI-50) at Week 4.The EASI will be assessed at every study visit. It quantifies the severity of a patient's atopic dermatitis based on both lesion severity and the percent of body surface area affected. The EASI is a composite score ranging from 0-72 that takes into account the degree of erythema, induration/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body regions, with adjustment for the percent of BSA involved for each body region and for the proportion of the body region relative to the whole body.
Efficacy - Peak Pruritus Numeric Rating Scale (NRS) | 28 days
  Efficacy will be assessed as change from Baseline to Week 4 in peak pruritus as measured with the 24-hour Peak Pruritus Numeric Rating Scale (NRS). Peak Pruitus NRS will be measured at each visit. The assessment consists of a patient-rated scale of 0-10, where 0 is "No itch" and 10 is the "Worst itch possible."
Efficacy - Whole body surface area (BSA) affected | 28 days
  This exploratory endpoint will be evaluated as the change in total score from Baseline at all visits in whole body BSA (body surface area) affected. Whole body BSA affected will be assessed at every visit.

SECONDARY OUTCOMES:
Frequency and severity of adverse events (local and systemic) | 28 days
  Adverse events will be coded using the most current release of MedDRA® (Medical Dictionary for Regulatory Activities). The number and proportion of subjects with adverse events will be summarized by treatment, system organ class, and preferred term for all adverse events, all adverse events considered by the investigator to be related to study drug, all serious adverse events, and all adverse events leading to study drug discontinuation
Plasma concentrations of RVT-501 | 7 days
  PK samples will be collected only at the Week 1 visit in 2-11 year old patients. RVT-501 will be measured in plasma by validated assay to confirm exposure.These plasma concentrations will be listed by metabolite, subject, treatment, and time; and will be summarized by analyte and time.
Plasma concentrations of M11 metabolite | 7 days
  PK samples will be collected only at the Week 1 visit in 2-11 year old patients. The M11 metabolite will be measured in plasma by validated assay to confirm exposure. These plasma concentrations will be listed by metabolite, subject, treatment, and time; and will be summarized by metabolite, treatment and time.

CONTACTS AND LOCATIONS:
Overall Officials: James Lee, MD, PhD, Study Chair — Dermavant Sciences, Inc.
Locations (7):
- United States (5):
  - Dermavant Investigational Site, Los Angeles, California
  - Dermavant Investigational Site, Oklahoma City, Oklahoma
  - Dermavant Investigational Site, Portland, Oregon
  - Dermavant Investigational Site, Dallas, Texas
  - Dermavant Investigational Site, San Antonio, Texas
- Canada (2):
  - Dermavant Investigational Site, Surrey, British Columbia
  - Dermavant Investigational Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Dermavant Sciences Official Website — https://dermavant.com/